CLINICAL TRIAL: NCT01438827
Title: Avanz Phleum Pratense Maintenance Dose
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV-G-02; AV-G-02
Record Dates: First submitted 2011-09-13; First posted 2011-09-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Allergic Rhinoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Avanz Phleum pratense 15,000 SQ+ (Active Comparator)
  Interventions: Drug: Avanz Phleum pratense
- Avanz Phleum pratense 4,000 SQ+ (Active Comparator)
  Interventions: Drug: Avanz Phleum pratense
- Injection with no active grass component (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avanz Phleum pratense — Suspension for Injection, Every 6 weeks for one year
  Arms: Avanz Phleum pratense 15,000 SQ+; Avanz Phleum pratense 4,000 SQ+
Drug: Placebo — Suspension for Injection, Every 6 weeks for one year
  Arms: Injection with no active grass component

SUMMARY:
The purpose of the trial is to evaluate the efficacy of two dosing schedules of Avanz SQ+ (Standardised Quality) Phleum pratense compared to placebo in subjects with grass pollen induced allergic rhinoconjunctivitis with or without asthma.

ELIGIBILITY:
Inclusion Criteria:

* A history of grass pollen allergy
* Positive skin prick test to grass
* Positive Immunoglobulin E test to grass

Exclusion Criteria:

* Other allergies overlapping the grass pollen season
* Severe Asthma (defined as a Forced expiratory volume in 1 second (FEV1) below 70 % after adequate treatment)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Recording of rhinoconjunctivitis symptoms | Daily recordings during the grass pollen season 2012
Recording of symptomatic allergy medication use | Daily recordings during the grass pollen seasons 2012

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Kleine-Tebbe, PD Dr., Principal Investigator — Clinical Research Center for Dermatology, Allergy and Asthma
Locations (1):
- UntersuchungsZentrum für Dermatologie, Allergologie und Asthma, Berlin, State of Berlin, Germany